CLINICAL TRIAL: NCT02641626
Title: Randomized Study About the Efficacy of an Urgent Coronariography in Patients With a Non-diagnostic Electrocardiogram Following Out of Hospital Cardiac Arrest.
Brief Title: Coronariography in OUt of hosPital Cardiac arrEst
Acronym: COUPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Vall d'Hebron (Other); Hospital Arnau de Vilanova (Other); Hospital Universitari de Bellvitge (Other); Hospital General Universitario Gregorio Marañon (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario Virgen Macarena (Other); Hospital Universitario de Canarias (Other); Germans Trias i Pujol Hospital (Other); Complejo Hospitalario Universitario de Santiago (Other); Hospital Universitario Principe de Asturias (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital de Leon (Other Government)
Responsible Party: Principal Investigator, Ana Viana Tejedor, MD. PhD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COUPE
Record Dates: First submitted 2015-12-20; First posted 2015-12-29 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; survival; neurologic prognosis; coronariography; hypothermia
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Urgent Coronary Angiography (Experimental): Urgent Coronary Angiography: as soon as possible, when the patient is randomized.
  Interventions: Procedure: Urgent Coronary Angiography
- Deferred coronariography (Active Comparator): Deferred coronary angiography: after extubation if the patient has a good neurologic prognosis.
  Interventions: Procedure: Deferred Coronary Angiography

INTERVENTIONS:
Procedure: Urgent Coronary Angiography — Diagnostic test for the evaluation of the coronary vasculature.
  Arms: Urgent Coronary Angiography
Procedure: Deferred Coronary Angiography — Diagnostic test for the evaluation of the coronary vasculature.
  Arms: Deferred coronariography

SUMMARY:
Prospective, multicenter, randomized clinical trial. Survivors from an out-of-hospital cardiac arrest (OHCA) without ST segment elevation in their EKG will be recruited. Potentially non-cardiac etiology of the cardiac arrest will be ruled out prior to randomization. Primary goal (treatment): to evaluate the efficacy of urgent vs deferred coronary angiography in survivors from OHCA without ST-segment elevation in the EKG.

DETAILED DESCRIPTION:
Prospective, multicenter and randomized clinical trial. Survivors from Out-of-Hospital Cardiac Arrest (OHCA) who do not show ST elevation in their EKG will be recruited in the present study. Potentially non-cardiac ethiology of the cardiac arrest will be ruled out prior to randomization. Afterwards, patients will be randomized to emergent or deferred (performed before discharge) coronary angiography. Both groups will receive routine care in the Acute Cardiac Care Unit, including therapeutic hypothermia.

The randomization will be in a 1:1 ratio to urgent or deferred coronary angiography.

The main objective of the study is to compare the effectiveness of an urgent coronary angiography and angioplasty if necessary versus a deferred coronary angiography in survivors from OHCA who after recovery of spontaneous circulation do not fulfill criteria for ST-elevation myocardial infarction.

The primary efficacy endpoint is a composite of in-hospital survival and six-month survival free of severe dependence, which will be evaluated by using the Cerebral Performance Category (CPC) Scale, being good prognosis represented by the categories 1 and 2.The safety endpoint will be a composite of MACE (Major Adverse Cardiac Events) including: death, reinfarction, bleeding or ventricular arrhythmias.

A total of 166 patients will be included. The estimated duration will be 42 months, with a target follow-up of 6 months. Periods will be divided as follows:

* Inclusion Period (selection of the population and data collection): 36 months.
* Monitoring, data analysis, statistical and clinical report: 6 months.

ELIGIBILITY:
Inclusion Criteria: survivors from out of hospital cardiac arrest who meet all the following criteria:

* Remain comatose after recovery of spontaneous circulation (ROSC) (Glasgow Coma Scale score equal or less than 8).
* Show a non-diagnostic electrocardiogram after ROSC (neither ST segment elevation nor left bundle branch block).
* Prior rule out of an obvious non-cardiac cause of the cardiac arrest (head CT scan and transthoracic echocardiogram).
* Absence of exclusion criteria.

Exclusion Criteria:

* Age <18 years.
* Pregnant women or women of childbearing age unless they have a negative pregnancy test.
* Time to return of spontaneous circulation longer than 60 minutes.
* Non-cardiac etiology of the comatose state: drug overdose, head injury or stroke.
* Acute myocardial infarction with ST segment elevation or left bundle branch block, because in those patients emergent angiography is mandatory.
* Hemodynamic instability (refractory cardiogenic shock despite vasoactive drugs or refractory arrhythmias), because in those patients an emergent angiography is mandatory.
* Known coagulopathy or bleeding.
* Refusal to participate in the study by the next of kin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Survival with good neurological outcome for activities of daily living (CPC 1-2). | 30 days.
  Survival with good neurological outcome for activities of daily living (CPC 1-2).
Survival with good neurological outcome for activities of daily living (CPC 1-2). | 6 months.
  Survival with good neurological outcome for activities of daily living (CPC 1-2).
MACE: death, myocardial infarction, clinically evident bleeding (BARC> 2) or ventricular arrhythmias. | 30 days.
  MACE: death, myocardial infarction, clinically evident bleeding (BARC> 2) or ventricular arrhythmias.
MACE: death, myocardial infarction, clinically evident bleeding (BARC> 2) or ventricular arrhythmias. | 6 months.
  MACE: death, myocardial infarction, clinically evident bleeding (BARC> 2) or ventricular arrhythmias.

SECONDARY OUTCOMES:
Hospital survival. | 30 days.
  Hospital survival.
Hospital survival. | 6 months.
  Hospital survival.
Neurological outcome assessed by the Cerebral Performance Category (CPC) Scale. | 30 days.
  Neurological outcome assessed by the Cerebral Performance Category (CPC)
Neurological outcome assessed by the Cerebral Performance Category (CPC) Scale. | 6 months.
  Neurological outcome assessed by the Cerebral Performance Category (CPC)
Left ventricular ejection fraction. | 30 days.
  Left ventricular ejection fraction.
Left ventricular ejection fraction. | 6 months.
  Left ventricular ejection fraction.
Infarction size | 30 days.
  Defined by the maximum CPK (creatine phosphokinase) and Troponin.
Vascular complications. | 30 days.
  Vascular complications such as pseudoaneurysms, arteriovenous fistulas, etc
Clinically evident haemorrhagia: BARC> 2 | 30 days.
  Clinically evident haemorrhagia: BARC> 2
Sustained ventricular arrythmias or requirement of cardioversion. | 30 days.
  Sustained ventricular arrythmias or requirement of cardioversion.
Renal impairment. | 30 days.
  A 50% increase of serum creatinine over a baseline level or an increase of >0.5 mg/dl
Reinfarction. | 30 days.
  According to the Universal Definition of Acute Myocardial Infarction
Stent Thrombosis | 30 days.
  Defined by the Academic Research Consortium (ARC).
Infections. | 30 days.
  Infections.
Length of intubation. | 30 days.
  Length of intubation.
Length of hospital stay. | 6 months.
  Length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Viana Tejedor, MD, PhD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

REFERENCES:
- [Result] Camuglia AC, Randhawa VK, Lavi S, Walters DL. Cardiac catheterization is associated with superior outcomes for survivors of out of hospital cardiac arrest: review and meta-analysis. Resuscitation. 2014 Nov;85(11):1533-40. doi: 10.1016/j.resuscitation.2014.08.025. Epub 2014 Sep 4. PMID 25195073
- [Result] Morrison LJ, Neumar RW, Zimmerman JL, Link MS, Newby LK, McMullan PW Jr, Hoek TV, Halverson CC, Doering L, Peberdy MA, Edelson DP; American Heart Association Emergency Cardiovascular Care Committee, Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on P. Strategies for improving survival after in-hospital cardiac arrest in the United States: 2013 consensus recommendations: a consensus statement from the American Heart Association. Circulation. 2013 Apr 9;127(14):1538-63. doi: 10.1161/CIR.0b013e31828b2770. Epub 2013 Mar 11. No abstract available. PMID 23479672
- [Derived] Viana-Tejedor A, Andrea-Riba R, Scardino C, Ariza-Sole A, Baneras J, Garcia-Garcia C, Jimenez Mena M, Vila M, Martinez-Selles M, Pastor G, Garcia Acuna JM, Loma-Osorio P, Garcia Rubira JC, Jorge Perez P, Pastor P, Ferrera C, Noriega FJ, Perez Macias N, Fernandez-Ortiz A, Perez-Villacastin J; COUPE Investigators. Coronary angiography in patients without ST-segment elevation following out-of-hospital cardiac arrest. COUPE clinical trial. Rev Esp Cardiol (Engl Ed). 2023 Feb;76(2):94-102. doi: 10.1016/j.rec.2022.05.013. Epub 2022 Jun 22. English, Spanish. PMID 35750580